CLINICAL TRIAL: NCT02246660
Title: RESveratrol To Improve Outcomes in oldeR pEople With PAD (the RESTORE Trial)
Acronym: RESTORE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mary McDermott, Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R21AG047510-01 (NIH); R21AG047510 (NIH)
Record Dates: First submitted 2014-09-18; First posted 2014-09-23 (Estimated); Results first posted 2018-04-30 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2017-11

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Artery Disease; Peripheral Arterial Disease; PAD
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Resveratrol - 500 mg/day (Active Comparator): The dose of Resveratrol will be 500 mg daily for six months. Resveratrol is taken orally. Resveratrol is a natural plant derivative.
  Interventions: Drug: Resveratrol
- Resveratrol - 125 mg/day (Active Comparator): The dose of Resveratrol will be 125 mg daily for six months. Resveratrol is taken orally. Resveratrol is a natural plant derivative.
  Interventions: Drug: Resveratrol
- Placebo (Placebo Comparator): Placebo will be taken orally for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Resveratrol — The dose of Resveratrol will be 500 mg daily for six months. Resveratrol is taken orally. Resveratrol is a natural plant derivative.
  OR
  The dose of Resveratrol will be 125 mg daily for six months. Resveratrol is taken orally. Resveratrol is a natural plant derivative.
  Other Names: Polygonum cuspidatum
  Arms: Resveratrol - 125 mg/day; Resveratrol - 500 mg/day
Drug: Placebo — Placebo will be taken orally for 6 months.
  Other Names: No active study medication
  Arms: Placebo

SUMMARY:
The RESTORE trial will determine whether resveratrol supplementation can improve walking performance in older people with lower extremity peripheral arterial disease (PAD). Resveratrol, a polyphenol and natural supplement, specifically targets several impairments associated with walking difficulty and mobility loss in people with PAD.

DETAILED DESCRIPTION:
Eight million men and women in the United States have lower extremity peripheral arterial disease (PAD). PAD is expected to be increasingly common as the population survives longer with chronic disease. Patients with PAD have greater functional impairment and faster functional decline compared to those without PAD. However, currently there are only two FDA approved medications for improving functional performance in patients with PAD. Furthermore, these FDA approved medications are only modestly beneficial for improving walking performance in patients with PAD.

Emerging evidence, including our pilot data, demonstrates that calf skeletal muscle mitochondria dysfunction contributes to functional impairment in people with PAD. Resveratrol, a polyphenol and natural supplement, has pharmacological properties that target specific mitochondrial impairments that are associated with functional impairment in older people with PAD. Animal models and preliminary human evidence show that resveratrol protects against ischemia-reperfusion injury, reduces inflammation, and improves endothelial dysfunction. Ischemia-reperfusion injury, inflammation, and endothelial dysfunction are all present in people with PAD and contribute to adverse outcomes in PAD.

We now propose a pilot study of 66 PAD participants age 65 and older: a double-blind, randomized controlled pilot clinical trial to provide preliminary data to address our hypothesis that resveratrol significantly improves lower extremity functioning in people with PAD by improving calf skeletal muscle oxidative metabolism, increasing calf skeletal muscle mitochondrial biogenesis, and improving systemic endothelial function in older people with PAD.

In our primary specific aims, we will determine 1) whether PAD participants randomized to resveratrol 500 mgs daily achieve greater increases or have less decline in six-minute walk performance at 6-month follow-up, compared to those randomized to placebo and 2) whether PAD participants randomized to resveratrol 125 mgs daily achieve greater increases or have less decline in six-minute walk performance at 6-month follow-up, compared to those randomized to placebo. In our secondary aims, we will determine whether PAD participants randomized to resveratrol have improved treadmill walking performance, increased calf muscle biopsy-measured mitochondrial function, increased calf muscle biopsy-measured mitochondrial biogenesis, and improved brachial artery flow-mediated dilation at six-month follow-up, compared to those randomized to control. For each secondary specific aim, participants randomized to 500 mgs of resveratrol (N=22) will be compared to those randomized to placebo (N=20) and participants randomized to 125 mgs of resveratrol (N=22) will be compared to those randomized to placebo (N=22), respectively. In an exploratory specific aim, we will determine whether participants randomized to resveratrol 125 mgs (N=22) have greater improvement in each study outcome compared to those randomized to resveratrol 500 mgs (N=22).

If our hypotheses are correct, results will be used to design a large, definitive randomized controlled trial of resveratrol therapy to improve lower extremity functioning and prevent mobility loss in the large and growing number of older people who are disabled by PAD. By studying two doses of resveratrol, our results will also provide guidance on the most optimal dose of resveratrol to use in a large definitive trial.

ELIGIBILITY:
Inclusion Criteria:

* Ankle-brachial index (ABI) < 0.90 at baseline screening (at visit), or, medical evidence of prior lower extremity revascularization if ABI ≥ 0.90.
* 65 or older

Exclusion Criteria:

* Above/below-knee amputation, critical limb ischemia, wheelchair-bound, or require the use of a walker or cane
* Other symptom(s) limiting walking ability, other than PAD
* Underwent/experienced lower extremity revascularization, a cardiovascular event, or coronary artery bypass surgery within 3 months of screening. Underwent major orthopedic surgery within 6 months of screening. Planning to have revascularization or major elective surgery within the next 6 months.
* Major medical illness including renal disease that requires dialysis or lung disease that requires oxygen
* Score of < 23 on Mini-Mental Status Examination at screening or major psychiatric illness
* Currently participating in a separate clinical trial
* Significant renal or liver dysfunction at baseline
* Does not successfully complete the study run-in period
* Has an extreme baseline 6 minute walk value (< 500 ft or > 1,600 feet )
* Treated for cancer during the last 2 years (unless prognosis is excellent)
* Severe hearing impairment or other communication difficulties (e.g. non-English speaking) or legally blind
* Diagnosis of Parkinson's disease
* Unable to return to medical center at required visit frequency
* Otherwise poorly suited to intervention (at the discretion of the PI)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary M McDermott, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gonzalez-Freire M, Moore AZ, Peterson CA, Kosmac K, McDermott MM, Sufit RL, Guralnik JM, Polonsky T, Tian L, Kibbe MR, Criqui MH, Li L, Leeuwenburgh C, Ferrucci L. Associations of Peripheral Artery Disease With Calf Skeletal Muscle Mitochondrial DNA Heteroplasmy. J Am Heart Assoc. 2020 Apr 7;9(7):e015197. doi: 10.1161/JAHA.119.015197. Epub 2020 Mar 21. PMID 32200714
- [Derived] McDermott MM, Peterson CA, Sufit R, Ferrucci L, Guralnik JM, Kibbe MR, Polonsky TS, Tian L, Criqui MH, Zhao L, Stein JH, Li L, Leeuwenburgh C. Peripheral artery disease, calf skeletal muscle mitochondrial DNA copy number, and functional performance. Vasc Med. 2018 Aug;23(4):340-348. doi: 10.1177/1358863X18765667. Epub 2018 May 8. PMID 29734865
- [Derived] McDermott MM, Leeuwenburgh C, Guralnik JM, Tian L, Sufit R, Zhao L, Criqui MH, Kibbe MR, Stein JH, Lloyd-Jones D, Anton SD, Polonsky TS, Gao Y, de Cabo R, Ferrucci L. Effect of Resveratrol on Walking Performance in Older People With Peripheral Artery Disease: The RESTORE Randomized Clinical Trial. JAMA Cardiol. 2017 Aug 1;2(8):902-907. doi: 10.1001/jamacardio.2017.0538. PMID 28403379

RESULTS

PARTICIPANT FLOW:
Groups:
- Resveratrol - 500 mg/Day: The dose of Resveratrol will be 500 mg daily for six months. Resveratrol is taken orally. Resveratrol is a natural plant derivative.
  Resveratrol: The dose of Resveratrol will be 500 mg daily for six months. Resveratrol is taken orally. Resveratrol is a natural plant derivative.
  OR
  The dose of Resveratrol will be 125 mg daily for six months. Resveratrol is taken orally. Resveratrol is a natural plant derivative.
- Resveratrol - 125 mg/Day: The dose of Resveratrol will be 125 mg daily for six months. Resveratrol is taken orally. Resveratrol is a natural plant derivative.
  Resveratrol: The dose of Resveratrol will be 500 mg daily for six months. Resveratrol is taken orally. Resveratrol is a natural plant derivative.
  OR
  The dose of Resveratrol will be 125 mg daily for six months. Resveratrol is taken orally. Resveratrol is a natural plant derivative.
Period: Overall Study
Arm/Group | Resveratrol - 500 mg/Day | Resveratrol - 125 mg/Day | Placebo
Started | 23 | 21 | 22
Completed | 23 | 20 | 21
Not Completed | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resveratrol - 500 mg/Day | Resveratrol - 125 mg/Day | Placebo | Total
Number analyzed (Participants) | 23 | 21 | 22 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.6 (7.3) | 73.6 (6.6) | 74.1 (6.1) | 74.4 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 7 | 21
  Male | 17 | 13 | 15 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 14 | 11 | 33
  White | 14 | 7 | 10 | 31
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Ankle Brachial Index [Mean (Standard Deviation); unit: Ratio] — A handheld Doppler probe was used to measure systolic blood pressures in the right brachial, dorsalis pedis, and posterior tibial arteries and left dorsalis pedis, posterior tibial, and brachial arteries. The ABI was calculated by dividing mean pressures in each leg by the mean of the 4 brachial pressures. A normal ABI is between 1.10- 1.30. A value of < 0.90 is about 70% sensitive and highly specific for the presence of peripheral artery disease. Lower ABI values indicate more severe PAD.
  Ratio | 0.69 (0.23) | 0.68 (0.15) | 0.63 (0.13) | 0.67 (0.18)
Current Smoker [Count of Participants; unit: Participants] | 4 | 5 | 5 | 14
Former Smoker [Count of Participants; unit: Participants] | 13 | 14 | 15 | 42
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.6 (5.5) | 28.9 (5.4) | 31.2 (4.8) | 29.9 (5.3)
Myocardial Infarction [Count of Participants; unit: Participants] | 1 | 1 | 0 | 2
Heart Failure [Count of Participants; unit: Participants] | 0 | 2 | 4 | 6
Stroke [Count of Participants; unit: Participants] | 3 | 6 | 0 | 9
Angina [Count of Participants; unit: Participants] | 2 | 1 | 4 | 7
Pulmonary Disease [Count of Participants; unit: Participants] | 5 | 3 | 2 | 10
Cancer [Count of Participants; unit: Participants] | 9 | 3 | 5 | 17
Diabetes [Count of Participants; unit: Participants] | 7 | 5 | 14 | 26
Intermittent Claudication [Count of Participants; unit: Participants] — Intermittent claudication was defined as exertional calf pain that did not begin at rest, caused the participant to stop walking, and resolved within 10 minutes of rest. Participants without intermittent claudication were either asymptomatic (ie, reported no exertional leg symptoms) or had exertional leg symptoms that did not meet criteria for intermittent claudication.
  Participants | 4 | 6 | 7 | 17
Exertional leg symptoms not consistent with classical intermittent claudication [Count of Participants; unit: Participants] | 14 | 12 | 11 | 37
Asymptomatic [Count of Participants; unit: Participants] | 5 | 3 | 4 | 12
6-Minute Walk Distance [Mean (Standard Deviation); unit: meters] | 357 (58) | 370 (65) | 354 (70) | 360 (63)
Total Treadmill Distance [Mean (Standard Deviation); unit: meters] | 529.4 (268.6) | 492.8 (261.2) | 443.3 (242.4) | 488.4 (255.9)
Treadmill distance at onset of leg symptom [Mean (Standard Deviation); unit: meters] | 271.1 (217.7) | 226.6 (123.4) | 218.0 (147.3) | 239.1 (168.5)
Cilostazol use [Count of Participants; unit: Participants] | 1 | 1 | 2 | 4
Pentoxifylline use [Count of Participants; unit: Participants] | 0 | 2 | 1 | 3
Antiplatelet therapy use [Count of Participants; unit: Participants] | 17 | 19 | 16 | 52
Statin use [Count of Participants; unit: Participants] | 14 | 16 | 17 | 47
Reported walking for exercise 3 or more times/week [Count of Participants; unit: Participants] | 9 | 4 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: 6-Minute Walk Distance, Meters
Description: Six month changes in 6-Minute Walk Distance (meters) in response to resveratrol therapy in patients with Peripheral Artery Disease were measured.
Time Frame: Baseline and 6 month follow-up
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Resveratrol - 500 mg/Day | Resveratrol - 125 mg/Day | Placebo
Number analyzed (Participants) | 23 | 20 | 21
meters | -12.8 (7.5) | 4.6 (8.1) | -12.3 (7.9)

ADVERSE EVENTS:
Arm/Group | Resveratrol - 500 mg/Day | Resveratrol - 125 mg/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/21 | 1/22
Serious Adverse Events (participants affected / at risk) | 4/23 | 0/21 | 4/22
Other Adverse Events (participants affected / at risk) | 19/23 | 18/21 | 15/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Resveratrol - 500 mg/Day (N=23) | Resveratrol - 125 mg/Day (N=21) | Placebo (N=22)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Allergy to lisinopril (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Toe amputation (Vascular disorders) | 0 | 0 (0) | 1 (1)
Urologic procedure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritic rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lower extremity revascularization (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Elective plastic surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Resveratrol - 500 mg/Day (N=23) | Resveratrol - 125 mg/Day (N=21) | Placebo (N=22)
Leg pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2
Foot pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Hand cramp (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Swelling (General disorders) | 1 | 1 | 2
Walking difficulty (General disorders) | 1 | 0 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Fever (Infections and infestations) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dizziness/headache (Nervous system disorders) | 2 | 0 | 0
Black stool (Gastrointestinal disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Weight loss (Metabolism and nutrition disorders) | 1 | 0 | 0
Nausea/vomiting (Gastrointestinal disorders) | 6 | 4 | 2
Diarrhea (Gastrointestinal disorders) | 14 | 7 | 11
Abdominal discomfort (General disorders) | 12 | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No